CLINICAL TRIAL: NCT05284448
Title: Effectiveness and Safety of Pentoxifylline in Treatment of Patients With Nonalcoholic Steatohepatitis
Brief Title: Pentoxifylline in Treatment of Patients With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, ahmed salah saad abomandour, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 312
Record Dates: First submitted 2022-02-16; First posted 2022-03-17 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Pentoxifylline

STUDY DESIGN:
Intervention Model Description: Clinical trial, parallel, randomized, prospective, controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pentoxifylline Group (Experimental): 25 patients will receive pentoxifylline (Trental SR®) 400 mg three times daily with their standard therapy for 6 months.
  Interventions: Drug: pentoxifylline (Trental SR®)
- Control Group (No Intervention): 25 patients will receive their standard therapy only

INTERVENTIONS:
Drug: pentoxifylline (Trental SR®) — 400 mg three times daily
  Arms: Pentoxifylline Group

SUMMARY:
The aim of the present study is to evaluate the efficacy and safety of pentoxifylline in the treatment of non-alcoholic steatohepatitis patients.

DETAILED DESCRIPTION:
Nonalcoholic steatohepatitis(NASH) is the progressive form of Non-alcoholic fatty liver disease (NAFLD), is characterized by hepatocellular damage, inflammation, and liver fibrosis that can progress to cirrhosis, in 25% of patients, NAFLD progresses to NASH, which increases the risk for the development of cirrhosis, liver failure, and hepatocellular carcinoma. In patients with NASH, liver fibrosis is the main determinant of mortality.

Pentoxifylline (PTX) is a xanthine derivative drug with a wide range of actions at the cellular and molecular level. PTX possess anti-inflammatory, antioxidant activities. PTX have potential role in improvement of NASH . Also, PTX inhibits a number of pro-inflammatory cytokines including interleukin-1, interleukin-6 and tumor necrosis factor (TNF-α ) which play an important role in the pathogenesis and progression of NASH.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18- 60 years old.
2. Both sexes
3. Patients who have nonalcoholic steatohepatitis (NASH) will be diagnosed by

   1. clinical examination (obese, high body mass index).
   2. radiological criteria of fatty liver (abdominal ultrasonography).
   3. laboratory investigation (elevated liver enzymes aspartate transaminase (AST), alanine transaminase (ALT).
4. The ability to give informed consent
5. Appropriate exclusion of other liver diseases

Exclusion Criteria:

1- Patients with other diagnosed chronic liver diseases as viral hepatitis, metabolic and genetic disorders as Hemochromatosis, Wilson disease, autoimmune hepatitis and drug induced liver disease as well as patients with recent infection and those who refused to be entitled in the study.

2. Patients will be excluded if they had a history of past excessive alcohol drinking for a period longer than 2 years at any time in the past 10 years.

3. Patients also will be excluded if they take medications known to cause steatosis or taking medications that have shown benefits in previous NASH pilot studies, including vitamin E, , thiazolidinedione, and alpha-glucosidase inhibitors.

4. Patients with a history of hypersensitivity to PTX or the methylxanthines (caffeine, theophylline, and theobromine) will be excluded, as well as those with a history of cerebral

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
improvement in liver aminotransferases(ALT and AST) | 6 months compared to the baseline
  Difference between last and first measurements
NAFLD fibrosis score (NFS) | 6 months compared to the baseline
  Change in NAFLD fibrosis score (NFS) (lower score means better outcome).

SECONDARY OUTCOMES:
The Aspartate (AST) to Platelet Ratio Index (APRI) score: | 6 months compared to the baseline
  Change in (APRI) score (lower score means better outcome).
The Fibrosis-4 (FIB-4) values: | 6 months compared to the baseline
  Change in (FIB-4) values (lower values means better outcome).
Serum Alkaline Phosphatase level (ALP) | 6 months compared to the baseline
  Change in ALP serum level as inflammatory markers of NASH
Serum Gamma-glutamyl Transferase level (GGT) | 6 months compared to the baseline
  Change in GGT serum level as inflammatory markers of NASH
Serum total and direct bilirubin. | 6 months compared to the baseline
  Change in levels of serum total and direct bilirubin.
Waist circumference | 6 months compared to the baseline
  Change in waist circumference
Change in anthropometric measures | 6 months compared to the baseline
  including BMI etc.
Lipid profile | 6 months compared to the baseline
  Change in serum lipids
Glycated hemoglobin (HbA1C) | 6 months compared to the baseline
  Change in HbA1C level for patients with T2DM
Fasting blood glucose level | 6 months compared to the baseline
  Change in fasting blood glucose for patients with T2DM
Drugs adverse events | 6 months compared to the baseline
  Assessment of safety by reporting any adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab Zalat, PhD, Study Chair — Professor and Head of Clinical Pharmacy Department, Faculty of Pharmacy, Al-Azhar University(Girls, Cairo); Adel Gaber Bakr, PhD, Study Director — Assistant Professor of Pharmacology and Toxicology, Al-Azhar University (Boys, Assiut); Ahmed ElGhandour, MD, Study Director — Assistant Professor of Internal Medicine and Gastroenterology, Faculty of Medicine, Ain-Shams University; ahmed abomandour, Demonstrator, Principal Investigator — Demonstrator of Clinical Pharmacy Department, Faculty of Pharmacy, Al-Azhar University (Boys, Assiut)
Locations (1):
- Internal medicine and hepatology outpatient clinic at Ain Shams University Hospital., Cairo, Egypt

REFERENCES:
- [Background] Leoncini L, Vindigni C, Megha T, Funto I, Pacenti L, Musaro M, Renieri A, Seri M, Anagnostopoulos J, Tosi P. Epstein-Barr virus and gastric cancer: data and unanswered questions. Int J Cancer. 1993 Apr 1;53(6):898-901. doi: 10.1002/ijc.2910530605. PMID 7682538
- [Background] Girolami A. Tentative and updated classification of factor X variants. Acta Haematol. 1986;75(1):58-9. doi: 10.1159/000206084. No abstract available. PMID 3088890